CLINICAL TRIAL: NCT07390760
Title: Effects of Remote Ischemic Conditioning (RIC) Combined With Balance Training on Spinal Reflex Modulation in Children With Cerebral Palsy
Brief Title: Remote Ischemic Conditioning and Spinal Reflex Modulation in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Swati Manoharrao Surkar, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMCIRB 25-000932
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Children With Cerebral Palsy
Keywords: Remote Ischemic Conditioning; Cerebral Palsy; Spinal Reflex Modulation; H-reflex; Balance Training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are masked to group assignment (RLIC vs. Sham conditioning)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Conditioning (RIC) (Experimental): RIC is achieved via blood pressure cuff inflation to at least 20 mmHg above systolic blood pressure to 200 mmHg on the thigh of more affected lower extremity. RIC involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation and requires 45 minutes. RIC is performed on visits 1 - 5.
  Interventions: Behavioral: Remote Ischemic Condtioning (RIC); Behavioral: Sham conditioning
- Sham conditioning (Sham Comparator): Sham conditioning is achieved via blood pressure cuff inflation to 25 mm Hg on the thigh of the more affected LE. Sham involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation and requires 45 minutes. Sham conditioning is performed on visits 1-5.
  Interventions: Behavioral: Sham conditioning; Behavioral: Balance training

INTERVENTIONS:
Behavioral: Remote Ischemic Condtioning (RIC) — See descriptions under arm/group descriptions. RIC is delivered for 5 intervention visits. Visits 1 is the baseline assessment and training visit, and visits 2-4 are RIC plus training visits, Visit 5 is training and post assessment visit.
  Arms: Remote Ischemic Conditioning (RIC)
Behavioral: Sham conditioning — See descriptions under arm/group descriptions. Sham conditioning is delivered for 5 intervention visits. Visits 1 is the baseline assessment visit, visits 2-5 are training visits, and visit 5 is training and post assessment visit.
Behavioral: Balance training — All participants will undergo training on a balance board, learning to hold the board level within the 5- degree horizontal range. Participants perform the balance task for 15, 30-second trials per day at visits 1-5.
  Arms: Sham conditioning

SUMMARY:
Remote ischemic conditioning (RIC) is a clinically feasible intervention involving brief, sublethal periods of ischemia followed by reperfusion that has been shown to enhance motor performance, strength, and balance when combined with training in healthy adults and individuals with neurological conditions. Although RIC is thought to influence neuroplasticity through neural, metabolic, and humoral pathways, its effects on spinal-level mechanisms remain poorly understood. Emerging evidence indicates that neuroplastic adaptations occur not only at the cortical level but also within the spinal cord. Moreover, altered spinal reflex excitability is associated with spasticity, balance impairments, and functional limitations in children with cerebral palsy (CP), yet the role of spinal reflex modulations in response to RIC and balance training remains under expplored in this population. Therefore, this study aims to investigate the effects of RIC combined with balance training on spinal reflex modulation in children with CP.

DETAILED DESCRIPTION:
Remote ischemic conditioning (RIC) is a clinically feasible, non-invasive intervention that involves brief, sublethal periods of ischemia followed by reperfusion and has been shown to improve motor performance, strength, and balance when combined with training in healthy adults and individuals with neurological conditions. Evidence from animal and human studies suggests that RIC exerts neuroprotective effects through multifactorial mechanisms involving neural, metabolic, vascular, and humoral pathways, with emerging data indicating the involvement of peripheral and spinal pathways. Neuroplasticity in response to training is known to occur not only at the cortical level but also within spinal neural circuits, where altered spinal reflex excitability is associated with spasticity, balance impairments, and poor functional outcomes in children with cerebral palsy (CP). While balance and locomotor training have been shown to reduce spinal reflex excitability in this population, the effects of RIC on spinal reflex modulation remain largely unexplored. The specific aims of this study are to determine whether 1) RIC combined with balance training modulates spinal reflex excitability, as reflected by H-reflex measures, and 2) to examine whether RIC combined with balance training leads to greater improvements in balance performance compared to sham conditioning combined with training in children with CP.

In this study, 16 children with cerebral palsy (ages 8-17 years) will be recruited. They will be randomly allocated into two groups: (A) RIC and (B) Sham. The study will consist of five consecutive visits. During Visit 1, participants will undergo baseline testing of the soleus H-reflex using a DS8R stimulator. After baseline testing, they will complete the first training session, which will include one session of conditioning combined with balance training (15 trials per session) on a stability trainer (Lafayette, IN). Visits 2 to 5 will each consist of one session of conditioning and balance training (second to fifth training sessions). During Visit 5, following the training session, post-testing of the H-reflex will be conducted. The average of the first five trials of balance training on Visit 1 will be used as the pre-test balance performance, and the average of the last five trials of balance training on Visit 5 will be used as the post-test balance performance. Conditioning will be administered to the more affected lower extremity (thigh), and a pulse oximeter will be placed on the toe for monitoring.

It is hypothesized that, compared to sham conditioning, remote ischemic conditioning combined with balance training will result in greater reductions in H-reflex excitability and greater improvements in balance performance in children with cerebral palsy. This study will help clarify whether RIC induces spinal reflex modulations when paired with balance training, reflecting spinal-level neuroplasticity in children with CP. These findings may advance understanding of the spinal mechanisms underlying the therapeutic benefits of RIC and support its translation as an adjunct intervention in pediatric neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with cerebral palsy (CP) between the ages 8-17 years
2. Gross motor function classification system levels I-III
3. Mainstream in school and has sufficient cognition to follow the experiment instructions

Exclusion Criteria:

Children with other developmental disabilities such as autism and developmental coordination disorders Children with cognitive deficits such as inability to understand and follow commands, substantially lower performance at grade level in school, and/or communication problems Children with balance disorders such as vestibular disorders, posterior fossa tumor etc.

Children with known cardiorespiratory dysfunctions Children with sickle cell disease Children who are receiving other adjunct therapies such as transcranial magnetic stimulation, transcranial direct current stimulation, or vagal nerve stimulation Presence of lower extremity condition, injury, or surgery within last three months which could compromise conditioning and training.

Participants who are pregnant.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in maximal H-reflex amplitude (Hmax) | [Time Frame: Baseline, Day 5]
  The maximal (peak) H-reflex amplitude will be determined from the recruitment (stimulus-response) curve. The Hmax amplitude provides an estimate of the number or proportion of motor neurons (MNs) activated from the total MN pool, reflecting spinal reflex modulations and spinal neuroplasticity.
Change in Hmax/ Mmax Ratio | [Time Frame: Baseline, Day 5]
  The maximal H-reflex and maximal M-wave amplitudes will be determined from the recruitment curve procedure. Calculating the Hmax/Mmax ratio is a standardization method used to reduce variability in H-reflex amplitude across participants. This provides a better basis for comparison and a more reliable estimate of changes in spinal reflex modulations between participants.

SECONDARY OUTCOMES:
Change in Balance Performance | [Time Frame: Baseline, Day 5]
  The average amount of time in seconds that a participant maintains the stability platform within ±5° of horizontal position during 15 trials of 30 seconds each. The total score will range between 0-30 seconds. Higher balance score indicates better balance performance. Greater average balance time indicates better balance performance.

CONTACTS AND LOCATIONS:
Overall Officials: Swati M Surkar, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on NIH figshare network and will be made available on request.
Supporting Information: ICF
Time Frame: After publishing the results of the study
Access Criteria: Data will be made available upon request to the principal investigator.